CLINICAL TRIAL: NCT05737966
Title: Evaluation of Case Management for First Episode Psychosis Using the PEPsy-CM Checklist
Acronym: CHECKLISTPEP
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Other Study IDs: LOCAL/2022/RP
Record Dates: First submitted 2022-12-22; First posted 2023-02-21 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: First Episode Psychosis
Keywords: first episode of psychosis assertive community treatment; early intervention in mental health; case management; assertive community treatment

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: evaluation of professional practices — Evaluation of professional practices : evaluation of the case management carried out in a program for early psychosis in France using a checklist according good practices guidelines

SUMMARY:
Psychotic disorders are often chronic conditions that lead to impaired functioning, quality of life and social integration. Current research and recommendations for good practice are moving towards early detection and intervention. It is recognized that this leads to better adherence, alliance to care and knowledge of pathology for the patient, especially in young patients. For more than a decade, early intervention services (EIS) are opened in France over an increasingly large territory. Still too few studies assess the impact of these structures in France. These EIS offer a multimodal intervention (social, professional, psychotherapeutic). The intervention of case managers (or care coordinators in french) seems to be the core of EIS. The case manager has a fundamental role in the process of recovery in coordinating each individual's treatment and ensuring continuity of care.

The PEPsy-CM study aims to evaluate the effectiveness on the relapse rate of a 3 year Program for Early Psychosis based on Case Management (PEPsy-CM) compared to TAU in a population of young people with a FEP.

A qualitative evaluation of case management practice in EIS seems essential to assess the impact of case managers under real conditions.

Based on the Australian Good Practice Recommendations (EPICC integrity tools) and the case management practice manuals, the PEPsy-CM check-list questionnaire was developed to evaluate the practice of case management in the EIS in France. This check-list contains different 35 items. The final score between 1(poor) to 5 (good) is established to determine the quality of the case management. Qualitative data are also collected during the interview with the participants.

ELIGIBILITY:
Inclusion Criteria:

* Professional working in an early intervention center treating first episodes of psychosis
* Professional involved in the organization/management of the center or practicing case management.

Exclusion Criteria:

* Professional not working in the early intervention center
* Professional working in the early intervention center but not having a role in the organization or management of the center or as case manager
* Professional who does not take charge of people who have had a first psychotic episode

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Professional working in an early intervention center treating first episodes of psychosis
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2023-02-01 (Actual); Primary Completion 2023-09-01 (Actual); Study Completion 2023-09-01 (Actual)

PRIMARY OUTCOMES:
conformity to TIDieR checklist in each center and for each case manager interviewed | 1 year
  TIDieR checklist Patient - Use of the case management manual (yes or no)
conformity to TIDieR checklist in each center and for each case manager interviewed | 1 year
  TIDieR checklist Patient - Use of specific and validated tools for Psychoeducation (yes or no)
conformity to TIDieR checklist in each center and for each case manager interviewed | 1 year
  TIDieR checklist Patient - Use of an information brochure on First Episode Psychosis (yes or no)
conformity to TIDieR checklist in each center and for each case manager interviewed | 1 year
  TIDieR checklist Patient - Use of specific and validated tools to support families (yes or no)
conformity to TIDieR checklist in each center and for each case manager interviewed | 1 year
  TIDieR checklist Patient - Use of specific and validated tools for Motivational Interviewing (yes or no)
conformity to TIDieR checklist in each center and for each case manager interviewed | 1 year
  TIDieR checklist Patient - Presence of Individualized Therapeutic Plan (ITP) supervision system (yes or no)
conformity to TIDieR checklist in each center and for each case manager interviewed | 1 year
  TIDieR checklist Patient - Use of Individualized Therapeutic Plan (ITP) supervision system (yes or no)

SECONDARY OUTCOMES:
description of the global organisation of each center | 1 year
  Number of staff by trade
description of their involvement in the early intervention center | 1 year
  number of years experience

CONTACTS AND LOCATIONS:
Locations (1):
- Schandrin, Nîmes, France